CLINICAL TRIAL: NCT00489866
Title: Aripiprazole Augmentation of Antidepressants in PTSD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Durham VA Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VA IRB#01163
Record Dates: First submitted 2007-06-20; First posted 2007-06-21 (Estimated); Results first posted 2012-03-28 (Estimated); Last update posted 2015-03-31 (Estimated); Status verified 2015-03

CONDITIONS: PTSD
Keywords: PTSD; Antidepressant; Aripiprazole; OEF; OIF
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Aripiprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Aripiprazole (Experimental)
  Interventions: Drug: Aripiprazole
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aripiprazole — Aripiprazole: 5 mg taken once a day orally for 2 weeks, then Aripiprazole: 5-10 mg taken once a day orally for 2 weeks, then Aripiprazole: 5-15 mg taken once a day orally for 2 weeks, then Aripiprazole: 5-20 mg taken once a day orally for 2 weeks
  Arms: Aripiprazole
Drug: Placebo — Same as active drug.
  Arms: Placebo

SUMMARY:
The proposed investigation will determine the therapeutic potential of aripiprazole augmentation to a stable antidepressant regimen for reducing posttraumatic stress disorder (PTSD) symptoms, cognitive symptoms, psychotic symptoms, and depressive symptoms in veterans with PTSD.

ELIGIBILITY:
Inclusion Criteria:

* Outpatient veterans with posttraumatic stress disorder (PTSD)
* Receiving treatment with an antidepressant at a stable dose for 4 weeks
* Male or female
* Ages 18-65 years old

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2007-03; Primary Completion 2008-09 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christine E Marx, MD, MA, Principal Investigator — Durham VAMC
Locations (1):
- Durham VAMC 508 Fulton Street, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited for participation from 4/07 through 12/08. The study was closed to enrollment on 12/08.
Pre-assignment Details: This was a randomized, placebo-controlled study.
Groups:
- Placebo: Identical to Aripiprazole
Period: Overall Study
Arm/Group | Aripiprazole | Placebo
Started | 7 | 7
Completed | 5 | 7
Not Completed | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aripiprazole | Placebo | Total
Number analyzed (Participants) | 7 | 7 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 7 | 14
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.49 (2.64) | 36.14 (5.52) | 33.81 (11.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 4 | 5
  Male | 6 | 3 | 9
Region of Enrollment [Number; unit: participants]
  United States | 7 | 7 | 14

OUTCOME MEASURES:

1. Primary Outcome: Clinician Administered PTSD Scale (CAPS)
Description: Mean change scores (Week 2 minus Week 6) in posttraumatic stress disorder symptoms. Scores may range from 0 (no symptoms) to 136 (severe symptoms; score of 136 is based on the first 17 CAPS items administered).
  A reduced CAPS score indicates a reduction in (improvement) PTSD symptoms, while an increase in CAPS score indicates an increase (worsening) in PTSD symptoms.
Time Frame: Week 2 and Week 6
Population: Analysis was intention to treat.
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- PTSD Symptoms Aripiprazole Treated Group; PTSD Symptoms Placebo Treated Group: The Clinician Administered PTSD Scale (CAPS) was used to measure changes in PTSD symptoms across the duration of the study.Mean change scores in posttraumatic stress disorder symptoms. Scores may range from 0 (no symptoms) to 136 (severe symptoms; score of 136 is based on the first 17 CAPS items administered). A reduced CAPS score indicates a reduction in (improvement) PTSD symptoms, while an increase in CAPS score indicates an increase (worsening) in PTSD symptoms.
Arm/Group | PTSD Symptoms Aripiprazole Treated Group | PTSD Symptoms Placebo Treated Group
Number analyzed (Participants) | 7 | 7
Units on a scale | 18.6 (24.28) | 9.58 (11.)

2. Primary Outcome: Brief Assessment of Cognition in Affective Disorders (BAC-A)
Description: The BACS includes brief assessments of executive functions, verbal fluency, attention, verbal memory, working memory and motor speed. Z-scores are calculated from composite scores. Higher z-scores are indicative of better cognitive performance, lower z-scores are indicative of lower cognitive performance. Range of z-scores anticipated to be between -3 and 3. Mean change scores from week 2 and week 6 (Week 2 minus Week 6).
Time Frame: Week 2 and Week 6
Measure: Mean (Standard Deviation); unit: Units on a Scale
Groups:
- Cognitive Symptoms Aripiprazole Treated Group; Cognitive Symptoms PlaceboTreated Group: The BACS includes brief assessments of executive functions, verbal fluency, attention, verbal memory, working memory and motor speed. Z-scores are calculated from composite scores. Higher z-scores are indicative of better cognitive performance, lower z-scores are indicative of lower cognitive performance. Range of z-scores anticipated to be between -3 and 3.
Arm/Group | Cognitive Symptoms Aripiprazole Treated Group | Cognitive Symptoms PlaceboTreated Group
Number analyzed (Participants) | 7 | 7
Units on a Scale | -0.41 (1.23) | -0.14 (0.56)

3. Primary Outcome: Positive and Negative Symptoms Scale (PANSS)
Description: The PANSS is a widely used measure with several subdomains, including positive symptoms, negative symptoms, and general psychopathology of schizophrenia. Lower scores are indicative of fewer symptoms; higher scores are indicative of more symptoms. Total PANSS scores range from 0-20.Mean change scores from Week 2 and Week 6 (Week 2 minus Week 6)
Time Frame: Week 2 and Week 6
Population: Analysis was Intention to Treat. Last Observation Carried Forward was the imputation technique utilized.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Groups:
- Psychotic Symptoms Aripiprazole Treated Group; Psychotic Symptoms Placebo Treated Group: The PANSS is a widely used measure with several subdomains, including positive symptoms, negative symptoms, and general psychopathology of schizophrenia. Lower scores are indicative of fewer symptoms; higher scores are indicative of more symptoms. Total PANSS scores range from 0-20.
Arm/Group | Psychotic Symptoms Aripiprazole Treated Group | Psychotic Symptoms Placebo Treated Group
Number analyzed (Participants) | 7 | 7
Units on a Scale | 2.57 (12.04) | -5.1 (7.31)

4. Secondary Outcome: Connor-Davidson Resilience Scale (CD-RISC)
Description: This scale measures resilience. Range of scores (0-100). A score of 0 is suggestive of no resilience, a score of 100 is suggestive of high level of resilience. Change scores calculated at Week 2 and Week 6 (Week 2 minus Week 6).
Time Frame: Week 2 and Week 6
Population: Analysis was Intention to Treat. Last Observation Carried Forward was the imputation technique utilized.
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Resilience Symptoms Aripiprazole Treated Group; Resilience Symptoms PlaceboTreated Group: This scale measures resilience. Range of scores (0-100). A score of 0 is suggestive of no resilience, a score of 100 is suggestive of high level of resilience.
Arm/Group | Resilience Symptoms Aripiprazole Treated Group | Resilience Symptoms PlaceboTreated Group
Number analyzed (Participants) | 7 | 7
Units on a scale | -3.00 (28.27) | -2.03 (7.79)

5. Secondary Outcome: Beck Depression Inventory, Second Edition (BDI-II)
Description: The Beck Depression Inventory-II (BDI) is a very sensitive and widely used instrument used to detect depressive symptoms. It consists of 21 items that assess the intensity of depression in both clinical and non-clinical subjects. Each item is a list of four statements arranged in increasing severity regarding a particular symptom of depression. Scores range from 0 to 63 (higher scores suggest higher levels of depression). Change scores were calculated from Week 2 and Week 6 scores (Week 2 minus Week 6).
Time Frame: Week 2 and Week 6
Population: Analysis was Intention to Treat. Last Observation Carried Forward was the imputation technique utilized.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Groups:
- Depression Symptoms Aripiprazole Treated Group; Depression Symptoms Placebo Treated Group: The Beck Depression Inventory-II (BDI) is a very sensitive and widely used instrument used to detect depressive symptoms. It consists of 21 items that assess the intensity of depression in both clinical and non-clinical subjects. Each item is a list of four statements arranged in increasing severity regarding a particular symptom of depression.
Arm/Group | Depression Symptoms Aripiprazole Treated Group | Depression Symptoms Placebo Treated Group
Number analyzed (Participants) | 7 | 7
Units on a Scale | 8.0 (19.66) | 2.28 (12.12)

ADVERSE EVENTS:
Arm/Group | Aripiprazole | Placebo
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 6/7 | 6/7
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aripiprazole (N=7) | Placebo (N=7)
Agitation (Psychiatric disorders) | 1 (1) | 1 (1)
Restlessness (Psychiatric disorders) | 2 (2) | 0 (0)
Increased Motor (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Decreased Motor Activity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Malaise (Psychiatric disorders) | 1 (1) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 2 (2)
Drowsiness (General disorders) | 2 (2) | 1 (1)
Cramps (General disorders) | 1 (1) | 3 (3)
Tremor (General disorders) | 0 (0) | 1 (1)
Vertigo (General disorders) | 1 (1) | 0 (0)
Syncope (General disorders) | 0 (0) | 1 (1)
Cold Extremity (General disorders) | 1 (1) | 0 (0)
Dry Mouth (General disorders) | 1 (1) | 2 (2)
Nasal Congestion (General disorders) | 0 (0) | 1 (1)
Blurred Vision (General disorders) | 2 (2) | 1 (1)
Constipation (General disorders) | 0 (0) | 1 (1)
Sweating (General disorders) | 0 (0) | 1 (1)
Nausea (General disorders) | 0 (0) | 4 (4)
Vomiting (General disorders) | 0 (0) | 1 (1)
Diarrhea (General disorders) | 0 (0) | 1 (1)
Menstrual Disturbance (General disorders) | 0 (0) | 2 (2)
Decreased Interest in Sex (General disorders) | 1 (1) | 1 (1)
Impaired sexual performance (General disorders) | 2 (2) | 1 (1)
Dermatological (General disorders) | 0 (0) | 1 (1)
Joint Pain/Stiffness (General disorders) | 1 (1) | 0 (0)
Join pain/stiffness (General disorders) | 1 (1) | 2 (2)
Decreased appetite (General disorders) | 0 (0) | 2 (2)
Increased appetite (General disorders) | 0 (0) | 1 (1)
Headache (General disorders) | 1 (1) | 2 (2)

LIMITATIONS AND CAVEATS:
One of the primary limitations of this pilot clinical trial is small sample size. Results of this study will clearly need to be replicated in a larger cohort.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes